CLINICAL TRIAL: NCT03536338
Title: Spinal Stimulation Sit-to-Stand Training After Spinal Cord Injury
Acronym: Stim2Stand
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University College, London (Other)
Collaborators: The Neurokinex Charitable Trust (Other); Inspire Foundation (Unknown); Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/0625
Record Dates: First submitted 2018-04-06; First posted 2018-05-24 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injuries
Keywords: Sit-to-stand; Spinal Stimulation; transcutaneous
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Purposefully sampled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Sit-to-stand training alone
  Interventions: Other: Sit-to-stand Training
- Treatment (Experimental): Sit-to-stand training combined with Spinal Stimulation
  Interventions: Other: Spinal Stimulation; Other: Sit-to-stand Training

INTERVENTIONS:
Other: Spinal Stimulation — transcutaneous electrical stimulation of the lumbar spinal cord during rehabilitation.
  Arms: Treatment
Other: Sit-to-stand Training — Rehabilitation of standing from a chair using the Keiser Rack

SUMMARY:
An injury to the spinal cord can be life altering: with a 'complete' injury, the affected individual is unable to move their legs at all and may become wheelchair-bound. While a 'complete' injury suggests that the cord was completely severed, it is actually more common for some connections in the spinal cord to remain after it is injured but, for some reason, they are inactive or sleeping.

Electrical stimulation applied to the skin surface at the lower back appears to 'wake up' these remaining connections, allowing some (previously unavailable) leg movements. The first time they had this spinal stimulation (SS), people with long-standing 'complete' spinal cord injuries became able to move their legs and, after several weeks of SS, these movements seemed to increase. They also noticed other changes taking place, including improvements in their bladder control.

SS has been shown to cause strong leg extension movements, and one person with SCI stood up with SS, using minimal support. SS for standing may assist people with SCI to carry out daily tasks at home, which would hugely benefit the SCI community.

In this study we will explore whether SS enables people with SCI to stand up and whether regular sit-to-stand training combined with SS improves; i) standing ability; ii) bladder control and; iii) well-being, in people with SCI.

Ten volunteers with SCI will carry out an 8-week sit-to-stand training programme. Training will be carried out 3 times/week at Neurokinex using their Keiser Power Rack. The volunteers will be randomly assigned either to the control (sit-to-stand only) or test (sit-to-stand plus SS) group. Measurements will be taken before and after the training programme to assess standing ability, bladder function, and well-being.

DETAILED DESCRIPTION:
Recruitment and Initial Assessment:

Participants will be recruited from London Spinal Cord injuries Centre (LSCIC) at the Royal National Orthopaedic Hospital (RNOH) and Neurokinex neurological rehabilitation centres where the 8-week (24-session) training intervention will be carried out. The study will also be advertised via relevant newsletters, bulletin boards, websites and mailing lists.

First Appointment (Visit 1 - 1 session at RNOH):

Each participant will attend an initial session at the RNOH in Stanmore, lasting one to two hours. Participants will be given the opportunity to ask questions about the study and informed consent to participate in the study will be taken.

Following this, we will perform some simple tests to check muscle response to stimulation without undue discomfort. Stimulating electrodes will be placed over the lower back and recording electrodes will be placed on lower limb muscles. The BCMA will then be completed: participants will be placed in the supine position and asked to perform a number of motor tasks in response to verbal cues (e.g. bring knee to chest). Stimulation will then be delivered in varying patterns (e.g. pulse width and frequency) and intensities (0mA to 100mA) and responses will be recorded from lower limb muscles. From this, optimal electrode position, and threshold level to stimulation will be defined. Trains of stimulation will then be applied at a range of frequencies (1-100Hz) and intensities 0mA to 100mA (or the highest intensity tolerated by the participant, whichever is lower). This will provide information on the pre-intervention ability of the participant. At the end of this session we will arrange with the participant a date for the next baseline session at the Neurokinex location most convenient for the participant to travel too.

Heart rate and blood pressure will be monitored intermittently during all stimulation procedures with a blood pressure monitor. This will be taken before beginning to record a baseline response and any significant rise in systolic and diastolic blood pressure greater than 20 mmHg systolic or 10 mmHg diastolic above baseline is an indication of autonomic dysreflexia (AD). If an event of AD occurs we will temporarily remove the stimulation until blood pressure returns to baseline. If this effect continues to occur this participant will be withdrawn from the study.

Baseline Session (Visit 2 - 1 session at Neurokinex):

During the baseline session, we will record measures of participant's ability to perform sit-to-stand onto force plates both with stimulation and without stimulation. Again, adhesive electrodes will be placed over the lower back and lower limb muscles and a small device called a goniometer will be positioned across the knee joint to measure its position. SS parameters (intensity, frequency) will be defined based on the results of the first appointment. Participants will then perform sit-to-stand with and without stimulation. This will be performed using the Keiser Power Rack: a device that assists transferring in the sit-to-stand manoeuvre by partially supporting your bodyweight. During the SS testing, stimulation will be delivered during each transition from the seated position to standing, maintained during standing for approximately 4-5 minutes (with intensity reduced if required for comfort) and switched off during sit-down for approximately 2-3 minutes. Training will last for 45 mins (including application of harness & electrodes 1 hour). A neurological assessment using the ASIA Impairment Scale (AIS) will also be performed and participants will be asked to complete questionnaires/forms to assess your well-being, independence and bladder function following the session.

Optionally, the patient's recent clinical urodynamics results will be obtained from RNOH.

Training (Visits 3-26; 24 sessions (3days/week) at Neurokinex):

Participants will be purposively assigned to either the control (sit-to-stand training; n=5) or test (sit-to-stand training with spinal stimulation; n=5) group, based on the results of the baseline neurological assessment performed at the baseline session (ASIA; Appendix 11). An 8-week (24-session) training intervention will be carried out at Neurokinex (participants enrolled site) (http://www.neurokinex.org/). Each participant will be required to attend Neurokinex for training 3 times per week for 8 weeks; each session will last approximately one hour.

During each session:

* Participants will receive 40 minutes of sit-to-stand training using the Keiser Power Rack. With the amount of body weight assistance set to provide minimal assistance, and will be adjusted as necessary throughout training.
* Nintendo Wii Balance Boards will also be positioned under each foot to measure loading during stance and two load cells will read the amount of force offset by the grip bar whilst transferring/standing.
* Five sit-to-stands will be completed in each session, as follows: transfer from sit-to-stand, 4-5 mins standing, transfer from stand to sit-down, 2-3 mins rest.

The test group will additionally receive SS during training. SS parameters (intensity, frequency) will be defined based on the results of the first appointment (see above), and will be modified during training as required. SS will be delivered during each transition from the seated position to standing, maintained during standing (with intensity reduced if required for comfort) and switched off during sit-down.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury for >1 year
* SCI level C5 -- T12
* Aged >18 years
* AIS A-D
* Unable to stand from a chair unaided

Exclusion Criteria:

* Cardiac pacemaker
* Any other musculoskeletal diagnosis affecting the lower limbs
* Pregnancy
* Complex regional pain syndrome
* Implanted metal or active device at electrode site (caudle to T9; e.g. screws, contraceptive coil)
* Spinal malignancy
* Uncontrolled autonomic dysreflexia
* Neurological degenerative diseases
* Peripheral nerve damage affecting the lower limbs
* Currently on any form of anti-spasticity treatment (e.g. Botox)
* Osteoporotic - bone density T score less than-2.5 (critical value).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Lower limb motor control (Electromyography) | Two hours
  Muscle activity and voluntary movement in the lower limbs

SECONDARY OUTCOMES:
Sit-to-stand performance | 30 mins
  Muscle activity and movement when standing from a chair
Health-related quality of life (QoL) | 1 hour
  Questionnaires
Bladder function (Urodynamics) | 2 hours
  Measuring bladder pressure during bladder filling

CONTACTS AND LOCATIONS:
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No